CLINICAL TRIAL: NCT05965947
Title: Medical Nutrition Therapy and Diet Quality Among Survivors of Brain Injury - The HOME Study (Healthy Options Made Easy): Telehealth Nutrition Sessions for People Living With Brain Injury
Brief Title: The HOME Study (Healthy Options Made Easy): Telehealth Nutrition Sessions for People Living With Brain Injury
Acronym: HOME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama, Tuscaloosa (Other)
Collaborators: Academy of Nutrition and Dietetics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22-11-6135
Record Dates: First submitted 2023-06-29; First posted 2023-07-28 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Brain Injuries
Keywords: brain injury; Medical Nutrition Therapy; Registered Dietitian; diet quality; Healthy Eating Index
MeSH Terms: conditions — Brain Injuries | interventions — Nutrition Therapy; Nutrition Assessment

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with an intervention group and a control group.
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor will be blinded to the group assignment of participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medical Nutrition Therapy (Experimental): The intervention group will be scheduled for three one-on-one sessions with a Registered Dietitian, where they will receive nutrition education and counseling. Sessions with the Registered Dietitian will include a review of the client's nutrition assessment data, development of problem list with the client, nutrition diagnosis, assessment of motivation to change, a discussion of barriers and facilitators, an intervention plan, goal setting, and monitoring and evaluation. Because individuals with brain injury may not do their own grocery shopping and meal preparation, caregivers will be encouraged to attend sessions. Checklists will be used to ensure treatment fidelity across participants and nutrition sessions. Sessions will be conducted by telehealth and will be recorded for fidelity checks and ongoing research team training. Sessions will be scheduled approximately 2 weeks apart.
  Interventions: Behavioral: Medical Nutrition Therapy
- Nutrition Handout Packet (No Intervention): The control group will receive a packet of nutrition education handouts from the MyPlate program found at USDA.gov. The handouts are publicly available and represent nutrition information that could be readily accessed by individuals who want to change their dietary habits, but do not have access to services from a Registered Dietitian.

INTERVENTIONS:
Behavioral: Medical Nutrition Therapy — One-on-one nutrition assessment, education, and counseling with a Registered Dietitian.
  Other Names: nutrition therapy, nutrition counseling, nutrition education
  Arms: Medical Nutrition Therapy

SUMMARY:
Brain injury is a leading cause of disability in the United States. When survivors of brain injury recover from the initial injury and return home to live in the community, they often face chronic health conditions that warrant nutrition therapy, such as diabetes, high blood pressure, high cholesterol, and overweight and obesity. Typically, these individuals do not receive nutrition counseling.

Thus, the purpose of this clinical trial is to compare changes in diet quality between community-dwelling individuals with a history of brain injury who receive three individualized nutrition therapy sessions versus handouts only.

Our research question is:

Can nutrition counseling improve dietary intake among this population?

Participants will complete a survey, participate in three days of dietary recalls via Zoom or telephone, and receive either three individualized nutrition counseling sessions with a Registered Dietitian or standard of care (handouts).

Researchers will compare the diets of the recipients of the nutrition counseling to a control group who receives nutrition handouts to see if nutrition sessions with a Registered Dietitian improve dietary intake.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the impact of providing nutrition therapy on diet among a cohort of community-dwelling individuals with a history of brain injury.

In this pre/post study, 134 participants with brain injury will be recruited and randomized to the control or intervention group. All participants will complete a standard set of nutrition-related questionnaires to assess weight status, co-morbid conditions, food security, stressors, stress-related eating, eating behaviors, and diet quality.

The control group will receive a packet of nutrition education materials. The intervention group will receive the packet and one-on-one nutrition counseling with a Registered Dietitian.

Follow-up data collection will include repeating the dietary recalls and questionnaires. This will allow for an evaluation of the impact of nutrition therapy on diet quality among community-dwelling individuals with brain injury.

Aim: Evaluate the effectiveness of providing nutrition therapy on diet quality and stress-related eating among a cohort of community-dwelling individuals with brain injury

• Ho: Individuals who receive three nutrition therapy sessions with a Registered Dietitian will have greater increases in Healthy Eating Index (HEI) scores than those who receive only handouts (current practice).

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* History of brain injury
* Live in Alabama
* Live at home in the community
* Have internet access to join Zoom sessions

Exclusion Criteria:

* Under 18 years of age
* No history of brain injury
* Lives outside of Alabama
* Currently in a hospital, rehabilitation facility, group home, or other location other than 'home'
* Pregnant or breastfeeding
* Not able/willing to participate based on the Decision-Making Capacity Assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2023-06-12 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in Diet Quality | Baseline and approximately 6 weeks later
  Diet quality is measured using the Healthy Eating Index Score, which ranges from 0-100. Higher scores indicate better diet quality. The score will be calculated at baseline and approximately 6 weeks later, and these timepoints will be used to calculate the change in diet quality over the study duration.

CONTACTS AND LOCATIONS:
Overall Officials: Joy W Douglas, PhD, Principal Investigator — The University of Alabama; Linda L Knol, PhD, Principal Investigator — The University of Alabama
Locations (1):
- The University of Alabama, Tuscaloosa, Alabama, United States

IPD SHARING:
Plan to Share IPD: No